CLINICAL TRIAL: NCT00619684
Title: A Phase II Study of Lenalidomide Following Allogeneic Stem Cell Transplant for Multiple Myeloma Patients Who Relapse or Have Disease Progression
Brief Title: Lenalidomide in Treating Patients With Progressive or Recurrent Multiple Myeloma After a Donor Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2161.00; NCI-2009-01592 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2161.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2008-02-20; First posted 2008-02-21 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2017-05-18 (Actual); Status verified 2015-09

CONDITIONS: Refractory Multiple Myeloma; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide

ARMS (1):
- Treatment (lenalidomide) (Experimental): Patients receive lenalidomide PO on days 1-21. Courses repeat every 28 days for 2 years or longer in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lenalidomide

INTERVENTIONS:
Drug: lenalidomide — Given PO
  Other Names: CC-5013; IMiD-1; Revlimid

SUMMARY:
This phase II trial studies how well lenalidomide works in treating patients with progressive or recurrent multiple myeloma after a donor stem cell transplant. Lenalidomide may stop the growth of multiple myeloma by blocking blood flow to the cancer. It may also stimulate the immune system in different ways and stop cancer cells from growing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate response of relapsed or progressive multiple myeloma to lenalidomide after allogeneic stem cell transplant.

II. Proportion of patients achieving a complete, partial or minor response.

SECONDARY OBJECTIVES:

I. Evaluate toxicity and tolerability of lenalidomide in this setting.

II. For patients with chronic graft-versus-host disease (GVHD), evaluate the response to lenalidomide.

III. Evaluate time to progression (TTP).

IV. Evaluate overall survival (OS).

OUTLINE:

Patients receive lenalidomide orally (PO) on days 1-21. Courses repeat every 28 days for 2 years or longer in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form
* Able to adhere to the study visit schedule and other protocol requirements
* Multiple myeloma, having undergone an allogeneic stem cell transplant from a matched or mismatched related or unrelated donor and have relapsed or have disease progression
* Relapse is defined as reappearance of monoclonal protein in serum or urine by immunofixation, new or increased bone lesions or hypercalcemia
* Disease progression is define as a 25% increase in monoclonal protein in serum or a 50% increase in 24 hour urinary monoclonal protein from the lowest level attained at any time point after allogeneic transplant or new or increased bone lesions or hypercalcemia
* All previous cancer therapy, including radiation, hormonal therapy and surgery, must have been discontinued at least 4 weeks prior to treatment in this study, excluding corticosteroids for GVHD
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2 at study entry
* Absolute neutrophil count >= 1.5 x 10^9/L
* Platelet count >= 50 x 10^9/L
* Serum creatinine =< 2.0 mg/dL
* Total bilirubin =< 1.5 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2 x upper limit of normal (ULN) or =< 5 x ULN if hepatic metastases are present
* Females of childbearing potential (FCBP) must adhere to the scheduled pregnancy testing as required in the Revlimid REMS™ program; FCBP must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 24 hours of prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide
* FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy
* Disease free of prior malignancies for >= 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast
* Able to take aspirin 81 or 325 mg daily as prophylactic anticoagulation (patients intolerant to acetylsalicylic acid [ASA] may use Coumadin or low molecular weight heparin)
* All study participants must be registered into the mandatory Revlimid REMS™ program, and be willing and able to comply with the requirements of Revlimid REMS™

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Pregnant or breast feeding females; (lactating females must agree not to breast feed while taking lenalidomide)
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Use of any other experimental drug or therapy within 28 days of baseline
* Known hypersensitivity to thalidomide
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
* Resistance to prior use of lenalidomide
* Concurrent use of other anti-cancer agents or treatments
* Known positive for human immunodeficiency virus (HIV) or infectious hepatitis, type A, B or C
* Acute GVHD grades 3 or 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-02; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Bensinger, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Lenalidomide)
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Lenalidomide)
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Response Rate, Defined as the Number of Patients Achieving Complete Response (CR), Partial Response (PR), or Minor Response (MR)
Description: CR: No Monoclonal Protein (MP) in the blood AND no serum/urine MP by Immunofixation (IF < 0) AND < 5% plasma cells in bone marrow aspirate.
  VGPR: More than 90% decrease of MP and urine M protein < 100 mg/d OR serum protein electrophoresis (SPEP)/urine protein electrophoresis(UPEP) negative but serum immunofixation (IFs) or IFu urine immunofixation (IFu) ) still positive.
  PR: Over 50% decrease of serum MP AND > 90% reduction in 24h urinary light chain excretion or M proteinuria < 200mg/d MR: Between 25 and 49% decrease of MP in the blood AND 50-89% reduction in 24h urinary light chain excretion (monoclonal proteinuria>200 mg/d)
Time Frame: Up to 9 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Lenalidomide)
Number analyzed (Participants) | 18
Participants
  Complete Response (CR) | 5
  Very Good Partial Response (VGPR) | 2
  Partial Response (PR) | 3
  Minimal Response (MR) | 1

2. Secondary Outcome: Adverse Events, Graded According to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0
Description: Grade 1-2 adverse events occurring in >10% of participants. Grade 3 or higher adverse events occurring in one or more participants.
Time Frame: Up to 30 days after completion of study treatment
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Lenalidomide)
Number analyzed (Participants) | 18
percentage of participants
  Grade 1-2 constipation | 28
  Grade 1-2 diarrhea | 17
  Grade 1-2 fatigue | 17
  Grade 1-2 myalgia | 17
  Grade 1-2 nausea | 11
  Grade 1-2 neuropathy | 11
  Grade 1-2 thrombocytopenia | 11
  Grade 3 pneumonia | 17
  Grade 3 H1N1 influenza | 11
  Grade 3 fever, hypoxia and neuropathy | 6
  Grade 3 myalgia | 6
  Grade 3 neuropathy | 6
  Grade 3 neutropenia | 44

3. Secondary Outcome: Number of Patients Requiring Dose Interruption, Dose Reduction or Discontinuance of Lenalidomide
Description: Dose interruption, dose reduction or discontinuation of lenalidomide due to toxicity, GVHD or disease progression
Time Frame: Up to 9 years
Population: Patients enrolled on the trial who received lenalidomide treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Lenalidomide)
Number analyzed (Participants) | 18
Participants | 13

4. Secondary Outcome: Number of Patients Who Experience Improvement in GVHD on Lenalidomide, Defined as the Reduction in Severity of GVHD as Defined by the National Institutes of Health (NIH) Consensus Criteria
Time Frame: Up to 9 years
Population: Patients who received lenalidomide on study
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Lenalidomide)
Number analyzed (Participants) | 18
Participants | 0

5. Secondary Outcome: TTP
Description: Time to Progression (TTP): Time from start of therapy to meeting the definition of Progressive Disease (PD).
  PD: 25% increase compared to the lowest value of:
  * Serum MP (absolute increase at least ≥ 0.5 g/dl)
  * Or: Urine MP (absolute increase at least > 200 mg/24h)
  * Or: for patients without measurable MP, Serum Free Light Chain test: the difference between involved and uninvolved FLC levels (absolute increase at least >100 mg/L)
Time Frame: Up to 9 years
Population: Patients who developed Progressive Disease while on lenalidomide treatment
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Lenalidomide)
Number analyzed (Participants) | 10
Months | 8.5 [1.2 to 43]

6. Secondary Outcome: Overall Survival
Description: Kaplan-Meier estimate of survival
Time Frame: At 1 and 2 years after starting treatment with lenalidomide
Population: Patients enrolled on trial who received lenalidomide therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Lenalidomide)
Number analyzed (Participants) | 18
percentage of participants
  Percent Overall Survival at 1 year | 71 [43 to 87]
  Percent Overall Survival at 2 years | 58 [31 to 78]

ADVERSE EVENTS:
Time Frame: Adverse event followed for 60 days after discontinuation of lenalidomide. Survival follow up up to 4 years.
Arm/Group | Treatment (Lenalidomide)
All-Cause Mortality (participants affected / at risk) | 8/18
Serious Adverse Events (participants affected / at risk) | 7/18
Other Adverse Events (participants affected / at risk) | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Lenalidomide) (N=18)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Influenza - H1N1 (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fever, hypoxia, neuralgia (General disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Lenalidomide) (N=18)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 3 (3)
Depression (Psychiatric disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5)
Peripheral neuropathy (Nervous system disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Fever (General disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Epistaxis (Ear and labyrinth disorders) | 1 (1)
Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Yeast infection (Infections and infestations) | 1 (1)
Skin tightness (Skin and subcutaneous tissue disorders) | 1 (1)
Jaw popping (Musculoskeletal and connective tissue disorders) | 1 (1)
Dry eyes (Eye disorders) | 1 (1)
Heartburn (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days